CLINICAL TRIAL: NCT04072094
Title: A Prospective Randomized Trial Comparing the Effect of Minimally Invasive Locking Plate Fixation and Reamed Intramedullary Nail Fixation on Patients With Gustilo I-III A Open Tibia Fracture
Brief Title: Minimally Invasive Locking Plate Fixation vs Reamed Intramedullary Nail Fixation on Patients With Open Tibia Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Taizhou Hospital (Other); Ningbo No.2 Hospital (Other); The First People's Hospital of Huzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: z2gk
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-08

CONDITIONS: Open tíbia Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Locking Plate Fixation (Experimental): Patients randomized to the Minimally Invasive Locking Plate Fixation arm will be treated with plate fixation. The plate may be applied in a percutaneous fashion. Any combination of locked and/or non-locked screws may be used.
  Interventions: Procedure: Minimally Invasive Locking Plate Fixation
- Intramedullary Nail Fixation (Active Comparator): Patients randomized to the Intramedullary Nail Fixation arm will be receive a standard locked intramedullary nail fixation. The nail must use at least one static interlock proximal to and one static interlock distal to the fracture site. The nail may be placed with a reamed technique.
  Interventions: Procedure: Intramedullary Nail Fixation

INTERVENTIONS:
Procedure: Minimally Invasive Locking Plate Fixation — Patients randomized to the Minimally Invasive Locking Plate Fixation arm will be treated with plate fixation. The plate may be applied in a percutaneous fashion. Any combination of locked and/or non-locked screws may be used.
  Other Names: Locking Plate Fixation
  Arms: Minimally Invasive Locking Plate Fixation
Procedure: Intramedullary Nail Fixation — Patients randomized to the Intramedullary Nail Fixation arm will be receive a standard locked intramedullary nail fixation. The nail must use at least one static interlock proximal to and one static interlock distal to the fracture site. The nail may be placed with a reamed technique.
  Arms: Intramedullary Nail Fixation

SUMMARY:
The best treatment for the open tibia fractures remains controversial. It is unknown whether minimally invasive locking plate or reamed intramedullary nail fixation will result in lower complication rates and better function.

DETAILED DESCRIPTION:
The best fixation method for open tibial fractures remains controversial. The current standard treatment options recommended the use of intramedullary nail for treating such fractures. Recent studies also showed favorable results for the use of plates in managing open tibial fractures. However, it is unknown whether locking plate or intramedullary nail fixation will result in lower complication rates and better function.

This study is a prospective, randomized trial to compare the safety and efficiency of minimally invasive plate osteosynthesis and reamed intramedullary nails in treating type I-II open tibial shaft fractures. The investigators hypothesize that neither intervention resulted in a superior disability rating at 12 months. Outcomes evaluated will include the rate of infection, the number of re-hospitalization for the complication, the time to bone healing, Patient-Reported outcome and quality of life and other complications.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 60 years inclusive
* Open diaphyseal fracture
* Gustilo-Anderson Type I, II, IIIA

Exclusion Criteria:

* Closed, periarticular or pathological fracture
* Gustilo-Anderson Type IIIB,IIIC
* Patients with concomitant fractures in the ipsilateral limb
* The patient is unable to medically tolerate general anesthesia
* The patient is unable to provide informed consent or comply with completing questionnaires
* Tibia already infected as diagnosed by a surgeon
* The patient has been diagnosed with a severe psychiatric condition

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
LEFS | 12 months
  failure.

SECONDARY OUTCOMES:
EQ-5D | 12 months
  Reported Outcome and Quality of Life

OTHER OUTCOMES:
SF-12 | 12 months
  Reported Outcome and Quality of Life
Fracture Healing | 12 months
  Fracture healing is measured by the treating surgeon using standard clinical criteria.
Complications | 12 months
  Soft tissue complications